CLINICAL TRIAL: NCT07373548
Title: Long-Term Clinical and Radiographic Outcomes Following Freehand and Guided Dental Implant Placement: A Randomized Controlled Trial Follow-Up
Acronym: SMART-ACCURACY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SmileDent Kft. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMP SMART 2224-4/2019
Record Dates: First submitted 2026-01-02; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Dental Implant; Edentulism; Navigation
Keywords: static guidance accuracy; dental implant; long-term follow-up

STUDY DESIGN:
Intervention Model Description: prospective, adaptive, parallel study with four arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- free hand (Experimental): free hand implant placement
  Interventions: Procedure: dental implant placement
- pilot (Experimental): pilot static guided implant placement
  Interventions: Procedure: dental implant placement
- partial (Experimental): partial static guided implant placement
  Interventions: Procedure: dental implant placement
- full (Experimental): full static guided implant placement
  Interventions: Procedure: dental implant placement

INTERVENTIONS:
Procedure: dental implant placement — placing dental implants

SUMMARY:
This study is a long-term clinical follow-up of a previously conducted randomized trial comparing different levels of surgical guidance in dental implant placement. The follow-up phase aims to evaluate peri-implant clinical and radiographic outcomes over an extended observation period of up to 67 months. Clinical parameters and marginal bone level changes are assessed to determine whether the accuracy benefits observed at implant placement translate into favorable long-term biological outcomes.

DETAILED DESCRIPTION:
The original clinical trial was designed to compare the accuracy of freehand and guided dental implant placement using different levels of surgical navigation. A total of 101 partially edentulous volunteers were enrolled and randomly assigned to one of four surgical protocols: freehand implantation, pilot-guided implantation, partially guided implantation, or fully guided implantation. Implant placement accuracy was evaluated by comparing the digitally planned implant positions with the actual postoperative implant positions using three-dimensional computerized analysis.

The present investigation represents an extended follow-up of this cohort, conducted to assess the long-term clinical performance of the placed implants. Follow-up evaluations began in February 2019 and continued until September 2024, resulting in a total observation period of up to 67 months. The extended duration exceeded the originally planned follow-up due to logistical interruptions related to the COVID-19 pandemic.

Clinical follow-up focused on peri-implant tissue health and marginal bone stability. Peri-implant probing depth was recorded as a clinical indicator of soft tissue conditions around the implants after delivery of the definitive prosthetic restorations. Measurements were performed at standardized sites around each implant, and mean probing depth values were calculated for longitudinal analysis.

Radiographic follow-up was performed using standardized bitewing radiographs to assess marginal bone levels. Marginal bone level was defined as the vertical distance between the implant platform and the alveolar crest, measured both mesially and distally. Because radiographic projection angles could not be fully standardized across all visits, individual calibration was performed for each implant using the known implant neck diameter provided by the manufacturer. This allowed reliable two-dimensional measurements despite variations in radiographic geometry.

The primary objective of this follow-up study is to describe long-term peri-implant clinical and radiographic outcomes following implant placement performed with varying levels of surgical guidance. Secondary objectives include assessing the stability of marginal bone levels over time and identifying potential differences between surgical protocols in long-term biological performance.

ELIGIBILITY:
Inclusion Criteria:

* • Age between 18 and 75 years

  * Partial edentulism in the maxilla or mandible involving 1-6 missing teeth, with no more than three adjacent missing teeth
  * Clinical conditions suitable for implant placement as assessed by the investigator or principal investigator (adequate bone and soft tissue conditions and acceptable occlusion)
  * Ability to communicate effectively with the investigators and willingness to comply with study procedures
  * Provision of written informed consent

Exclusion Criteria:

* • Pregnancy or breastfeeding

  * Women of childbearing potential without adequate contraception (for radiological safety reasons)
  * Conditions preventing safe intraoral manipulation (e.g., limited mouth opening, pronounced gag reflex)
  * Current or previous bisphosphonate therapy
  * History of radiotherapy involving the maxilla or mandible
  * International normalized ratio (INR) > 2.5
  * Known HIV, hepatitis B, or hepatitis C infection
  * Known allergy to any component of the implant or surgical guide system
  * Poor oral hygiene
  * Substance abuse
  * Smoking
  * Untreated periodontal disease
  * Any systemic disease or condition judged by the principal investigator to pose an unacceptable risk to the participant or to compromise study completion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2024-02-11 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Implant Survival | Up to 67 months post-implant placement
  Long-term survival of dental implants placed in the four study arms defined in the IMP SMART 002 trial, evaluated as a direct temporal extension of the IMP SMART 002 protocol (OGYÉI approval number 2224-4/2019). Implant survival is defined as the implant remaining in situ and functional without removal.

SECONDARY OUTCOMES:
Long-Term Tolerability and Safety | Up to 67 months post-implant placement
  Assessment of the long-term tolerability and safety of the implanted dental implants based on the occurrence of adverse events and complications.
Number of events of prosthodontic complications | From prosthetic delivery up to 67 months of follow-up
  Prosthodontic complications of the screw-retained implant-supported veneered zirconia prostheses in both arches were monitored and recorded throughout the 67-month follow-up period. Complications were calculated based on the occurrence of the following events: loss of access-hole cover, framework fracture, veneering ceramic fracture, prosthetic tooth fracture, abutment screw loosening, abutment screw fracture, prosthesis screw loosening, and prosthesis screw fracture.
Oral Health-Related Quality of Life Assessed by the OHIP-14 Questionnaire | Up to 67 months post-implant placement
  Patient-reported oral health-related quality of life assessed longitudinally using the validated Hungarian version of the Oral Health Impact Profile-14 (OHIP-14) questionnaire. The OHIP-14 evaluates the impact of dental implants and implant-supported prosthetic restorations on functional, physical, psychological, and social aspects of daily life.
  Measurement Tool: OHIP-14 questionnaire (14 items). Unit of Measure: Total OHIP-14 score (sum score ranging from 0 to 56), where higher scores indicate poorer oral health-related quality of life.
  Method of Assessment: For each visit, individual item scores (5-point Likert scale: 0 = never to 4 = very often) are summed to calculate a total OHIP-14 score. Mean total scores are calculated across the study population at each visit to evaluate changes in oral health-related quality of life over time.
Marginal Bone Loss | From prosthetic delivery up to 67 months of follow-up
  Long-term assessment of peri-implant marginal bone changes using standardized radiographic evaluation.
  Unit of Measure: Millimeters (mm)
Probing Depth | From prosthetic delivery up to 67 months of follow-up
  Long-term assessment of peri-implant soft tissue health by measuring probing depth around dental implants.
  Unit of Measure: Millimeters (mm)
Gingival Index | From prosthetic delivery up to 67 months of follow-up
  Long-term assessment of peri-implant gingival inflammation using the Gingival Index score.
  Unit of Measure: Score (Units on a Scale)
Plaque Index | From prosthetic delivery up to 67 months of follow-up
  Long-term assessment of oral hygiene status around dental implants using the Plaque Index score.
Width of Keratinized Gingiva | From prosthetic delivery up to 67 months of follow-up
  Long-term assessment of peri-implant soft tissue characteristics by measuring the width of keratinized gingiva.
  Unit of Measure: Millimeters (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Smile Dent, Szeged, Csongrád megye, Hungary